CLINICAL TRIAL: NCT04158518
Title: De-escalation of Chemoradiotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: De-escalation Protocols in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chaosu Hu (Other)
Responsible Party: Sponsor-Investigator, Chaosu Hu, Principal Investigator, Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019-NPC001
Record Dates: First submitted 2019-11-07; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; De-escalation
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toxicities reduced treatment (Experimental): Patients receive docetaxel(75mg/m2 d1) and cisplatin(25 mg/m2 d1-3) every 3 weeks for 3 cycles as induction chemotherapy, followed by omitting concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 50% Partial Response(PR).
  Interventions: Radiation: Toxicities reduced treatment
- Conventional treatment (Active Comparator): Patients receive docetaxel(75mg/m2 d1) and cisplatin(25 mg/m2 d1-3) every 3 weeks for 3 cycles as induction chemotherapy, followed by concurrent cisplatin chemotherapy with standard radiation dose when responses to induction chemotherapy are less than 50% Partial Response(PR).
  Interventions: Radiation: Conventional treatment

INTERVENTIONS:
Radiation: Toxicities reduced treatment — Drug: docetaxel and cisplatin (Induction chemotherapy) Patients receive docetaxel (75 mg/m2 d1) and cisplatin (25mg/m2 d1-3) every 3 weeks for 3 cycles before IMRT.
  Omitting concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 50% Partial Response(PR).
  Radiation: IMRT Intensity modulated-radiotherapy (IMRT) is given as 2.2 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 or 70.4 Gy to the primary tumor.
  Arms: Toxicities reduced treatment
Radiation: Conventional treatment — Drug: docetaxel and cisplatin (Induction chemotherapy) Patients receive docetaxel (75 mg/m2 d1) and cisplatin (25mg/m2 d1-3) every 3 weeks for 3 cycles before IMRT.
  Concurrent cisplatin chemoradiotherapy delivered when responses to induction chemotherapy are less than 50% Partial Response(PR).
  Radiation: IMRT Intensity modulated-radiotherapy (IMRT) is given as 2.2 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 or 70.4 Gy to the primary tumor.
  Arms: Conventional treatment

SUMMARY:
The purpose of this study is to explore the efficacy and safety of image guided de-escalation protocols in patients with locoregionally advanced nasopharyngeal carcinoma (NPC). So the investigators studied whether toxicities reducing treatment with omitted concurrent chemotherapy after good response to induction chemotherapy would maintain survival outcomes while improving tolerability for patients with locoregionally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of nasopharyngeal carcinoma
* Stage III or IVA according to UICC/AJCC 8th staging system
* Age ≥18
* No prior anti-tumor treatment
* Karnofsky Performance Score (KPS)≥70
* Adequate blood supply
* Informed consent obtained

Exclusion Criteria:

* Can not take contrast-MRI imaging
* Pregnant
* Combined with other malignant tumor (except basal cell carcinoma of skin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | 3 year
  Disease Free Survival

SECONDARY OUTCOMES:
OS | 3 year
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, MD, Principal Investigator — Fudan University Shanghai Cancer Centre
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, China